CLINICAL TRIAL: NCT06556303
Title: THE EFFECT OF ACUPRESSURE ON SLEEP QUALITY OF NURSING STUDENTS: A Randomised Controlled Study
Brief Title: Acupressure and Sleep Quality of Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Sibel Serce, Asst. Prof., University of Gaziantep
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 13082024
Record Dates: First submitted 2023-06-16; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Poor Quality Sleep
Keywords: Nursing students; Acupressure; Sleep quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental study model
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Comparison of Some Characteristics of the Students with Sleep Quality Mean Score (Experimental): The students in the intervention group were subjected to acupressure on the right and left sides of Shenmen (HT7) acupuncture point of the heart meridian, Sanyinjiao (SP6) acupuncture point of the spleen meridian, Neiguan (PC6) acupuncture point of the pericardium point, and Tian-Zhu (BL10) acupuncture point of the neck. The researcher having the certificate practised acupressure on each point for two minutes each, totalling 16 minutes, three days a week for four weeks.
  Interventions: Other: Acupressure
- Students and Their Sleep Quality Mean Score Before Acupressure Application (Experimental): The students in the intervention group were subjected to acupressure on the right and left sides of Shenmen (HT7) acupuncture point of the heart meridian, Sanyinjiao (SP6) acupuncture point of the spleen meridian, Neiguan (PC6) acupuncture point of the pericardium point, and Tian-Zhu (BL10) acupuncture point of the neck. The researcher having the certificate practised acupressure on each point for two minutes each, totalling 16 minutes, three days a week for four weeks.
  Interventions: Other: Acupressure
- Comparison of Sleep Quality Total Scores and Subscale Mean Scores of Intervention and Control Groups (Experimental): The students in the intervention group were subjected to acupressure on the right and left sides of Shenmen (HT7) acupuncture point of the heart meridian, Sanyinjiao (SP6) acupuncture point of the spleen meridian, Neiguan (PC6) acupuncture point of the pericardium point, and Tian-Zhu (BL10) acupuncture point of the neck. The researcher having the certificate practised acupressure on each point for two minutes each, totalling 16 minutes, three days a week for four weeks.
  Interventions: Other: Acupressure

INTERVENTIONS:
Other: Acupressure — Acupressure

SUMMARY:
This randomised, controlled and experimental study was conducted between 15 April and 15 June 2022 to examine the effect of acupressure on sleep quality of fourth-year nursing students. The population of the study consisted of all fourth-year nursing students and the sample consisted of 53 students who met the inclusion criteria. Approval from the ethics committee, permission from the institution and consents from the students were obtained before the research. The participants were assigned to intervention (n=26) and control (n=27) groups by simple random sampling method. The students in the intervention group were subjected to acupressure on the right and left sides of Shenmen (HT7) acupuncture point of the heart meridian, Sanyinjiao (SP6) acupuncture point of the spleen meridian, Neiguan (PC6) acupuncture point of the pericardium point, and Tian-Zhu (BL10) acupuncture point of the neck. The researcher having the certificate practised acupressure on each point for two minutes each, totalling 16 minutes, three days a week for four weeks. A questionnaire and the Pittsburgh Sleep Quality Index (PSQI) were applied at the beginning of the study, and the PSQI was applied again at the end of the fourth week. Total score of the PSQI ranges from 0 to 21. A total score higher than five indicates poor sleep quality. It was found that the PSQI total mean score of the intervention group dropped from 8.53±2.45 to 6.38±3.64, while the PSQI total mean score of the control group decreased from 9.40±1.62 to 8.40±3.48 (p<0.05). Also, subjective sleep quality, sleep disturbances and daytime dysfunction significantly decreased in the intervention group (p<0.05).

DETAILED DESCRIPTION:
Sleep is a brain function and is crucial for the maintenance of physical and mental health. Sleep, during which we spend approximately one-third of the life, is also a multidimensional and active state1. Therefore, it has been pointed out that sleep is a priority requirement in terms of protection and maintenance of health and quality of life2. In the literature, it is reported that the prevalence of sleep disorder is 5% in the world and 21.8% in Turkey, sleep-related complaints are frequently experienced, and poor sleep leads to physical and psychological disorders3. Quality sleep is described as a person who feels energetic and ready for a new day after waking up. Sleep quality includes quantitative aspects of sleep such as sleep latency, sleep duration and the number of wake-ups in a night, as well as subjective aspects such as the depth and restfulness of sleep. However, working conditions, occupational factors and stress can significantly affect the structure and quality of sleep. Sleeping disorders are observed more frequently, especially in patients with chronic diseases, healthcare personnel and people who work on call. The on-call working system of healthcare professionals disrupts the natural rhythm of human physiology and the sleep-wake cycle4. Studies have shown that the on-call system disrupts the natural circadian rhythm and may lead to serious changes in the gastrointestinal, cardiovascular and metabolic systems as well as the family and social life of nurses1. As known, the nursing profession, providing uninterrupted health care, requires working in shifts and may predispose to the appearance of sleeping disorders in this profession5. Also, an intensive and practical education programme is implemented during nursing education in Turkey and this may cause students to suffer from problems such as sleep deprivation, loss of performance and concentration6. A study conducted with nursing students found that students suffer from sleep problems more frequently compared to the general population and this causes physical problems and accidents as well as psychosocial problems such as low academic success, substance withdrawal, substance addiction, and emotional-behavioural and eating disorders7. However, it is very important that nursing students, who will deliver health services to society following their education, should have a complete physical and mental well-being and be able to maintain this state6. Accordingly, it is significant that students who are educated in health disciplines, all of whose practices are related to human health and therefore require an open mind and attention, acquire healthy lifestyle habits. Therefore, it is recommended to identify the present condition to ensure adequate and quality sleep, one of the parameters of a healthy lifestyle, and to use some supportive methods for enhancing the quality of sleep7. Today, pharmacological and non-pharmacological approaches are generally utilised to manage sleep disorders. However, non-pharmacological approaches may be preferred more due to their fewer side effects8. Acupressure, one of these methods, is stressed to be a reliable and effective practice that positively affects sleep by releasing neural mediators in order to enhance sleep quality9. Many studies have also found that acupressure practice has positive effects on sleep quality.10,11 Başer et al., found that acupressure applied on Tian-Zhu, Ju-Que, YongQuan, Bai-Hui and Nei-Guan points for 24 minutes three times a week for eight weeks in the elderly improved sleep quality.8,12 Similarly, it was found that acupressure applied on Neiguan (PC6), Shen Men (HT7), Sanyinjiao (SP6), Yintang (EX-HN3) and Tay (EX5) points for two minutes and once a day for two days improved sleep quality in patients who were followed for acute myocardial infarction.13 This information clearly suggests that acupressure contributes positively to sleep quality. Therefore, this study aimed to assess the effect of acupressure applied to the fourth-year nursing students who attended their practical education in clinics on sleep quality.

MATERIALS AND METHODS This randomised, controlled and experimental study was conducted between 15 April and 15 June 2022 to evaluate the effect of acupressure on fourth-year nursing students on sleep quality. The population of the study consisted of all fourth-year nursing students who continued their clinical practice education, and the sample consisted of 53 students with a PSQI score of five and above. The minimum sample size required in both groups to find the difference of 4.50 units (Cohen's d=1.45) between two mean scores between the acupressure group and the non-acupressure group in terms of Pittsburgh Sleep Quality Index (PSQI) scores to be significant was calculated as 12 (α=0.05, 1-β=0.90) (12). Students were assigned to intervention and control groups by using a computer programme for randomisation. The study included fourth-year nursing students of the relevant faculty, who had a PSQI score of five or above, had no comorbidities (heart disease, migraine, psychiatric comorbidities, etc.), were not on medication for sleep problems, and volunteered to participate in the study.14 The students who failed to meet the inclusion criteria were excluded from the study.

Acupressure Acupressure was applied on Shenmen (HT7)9,11 (Image 1),15 located at the tip of the ulnar bone and the heart meridian, Sanyinjiao (SP6) (Image 2),16 the sixth point of the splenic meridian approximately four fingers above the ankle, Neiguan (PC6) (Image 3),17 a pericardium point located between two tendons three fingers above the wrist in the forearm, and Tian-Zhu (BL10) (Image 4)18 acupuncture points on the neck of the students in the intervention group for two minutes on each point, on the right and left, for a total of 16 minutes, three days a week for four weeks. In both intervention and control groups, a questionnaire and the Pittsburgh Sleep Quality Index (PSQI) were applied at the beginning of the study, and the PSQI was applied again at the end of the fourth week.13 Acupressure was applied by the researcher having a certificate on the examination couch in a room prepared for the application by scheduling an appointment for each student. The student was placed in the Fowler position for the acupressure on Shenmen (HT7), Sanyinjiao (SP6) and Neiguan (PC6) points and in the supine position for the acupressure on Tian-Zhu (BL10) point. Any application was not practised in the control group. However, one session of acupressure was applied at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* The study included fourth-year nursing students of the relevant faculty, who had a PSQI score of five or above, had no comorbidities (heart disease, migraine, psychiatric comorbidities, etc.), were not on medication for sleep problems, and volunteered to participate in the study

Exclusion Criteria:

* The students who failed to meet the inclusion criteria were excluded from the study.

Ages: 19 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change in sleep during the Follow-up | one mounth
  This scale consists of seven subscales (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleep medication and daytime dysfunctions) and 19 items. The sum of all subscales is assessed with a total sleep quality score ranging from 0 to 21. A total score higher than five indicates poor sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Serçe, Asst. Prof., Principal Investigator — Gaziantep Universty; Ozlem Ovayolu, Prof, Study Chair — Gaziantep Universty; Nimet Ovayolu, Prof, Study Chair — SANKO Universty
Locations (1):
- Gaziantep Unıversty, Gaziantep, Sehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No